CLINICAL TRIAL: NCT03637361
Title: A Phase 1 Study to Investigate the Safety, Tolerability, and Pharmacokinetic Profile of Single Ascending Doses of REL-1017 (d-Methadone) in Healthy Subjects
Brief Title: Safety, Tolerability and Pharmacokinetics of Single Ascending Doses of REL-1017 (d-Methadone)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Relmada Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: REL-1017-111
Record Dates: First submitted 2018-08-10; First posted 2018-08-20 (Actual); Last update posted 2019-08-01 (Actual); Status verified 2018-08

CONDITIONS: Neuropathic Pain
MeSH Terms: conditions — Neuralgia | interventions — D-methadone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Arm 1 (Placebo Comparator): 100 mL Ocean Spray® Diet Cranberry Juice
  Interventions: Drug: Placebo
- Arm 2 (Experimental): REL-1017 5 mg in 100 mL of Ocean Spray® Diet Cranberry Juice
  Interventions: Drug: REL-1017
- Arm 3 (Experimental): REL-1017 20 mg in 100 mL of Ocean Spray® Diet Cranberry Juice
  Interventions: Drug: REL-1017
- Arm 4 (Experimental): REL-1017 60 mg in 100 mL of Ocean Spray® Diet Cranberry Juice
  Interventions: Drug: REL-1017
- Arm 5 (Experimental): REL-1017 100 mg in 100 mL of Ocean Spray® Diet Cranberry Juice
  Interventions: Drug: REL-1017
- Arm 6 (Experimental): REL-1017 150 mg in 100 mL of Ocean Spray® Diet Cranberry Juice
  Interventions: Drug: REL-1017

INTERVENTIONS:
Drug: REL-1017 — The investigational product, REL-1017 is prepared as a solution with Ocean Spray® Diet Cranberry Juice on site to obtain a final volume of 100 mL for dosing. The study drug will be administered as a solution of 5 mg, 20 mg, 60 mg, 100 mg, 150 mg or 200 mg REL-1017, based on randomization prepared in Ocean Spray® Diet Cranberry Juice with a final volume of 100 mL
  Other Names: (d-Methadone)
  Arms: Arm 2; Arm 3; Arm 4; Arm 5; Arm 6
Drug: Placebo
  Arms: Arm 1

SUMMARY:
This study evaluated the safety, tolerance, and pharmacokinetics (PK) of d-methadone in a limited dose range, in single administrations in humans.

DETAILED DESCRIPTION:
This was a phase 1, single-center study carried out in healthy male and female subjects to investigate the safety, tolerability, and PK of d-methadone. This was a double-blind, randomized, placebo-controlled study in 6 sequential cohorts of healthy subjects. Single oral doses of d-methadone were investigated in sequential cohorts. The proposed doses were 5 mg, 20 mg, 60 mg, 100 mg, 200 mg, 300 mg, and 400 mg. The decision to enroll the sequential cohort at the next dose level was based on the safety data and available PK data from previous doses. Dose escalation depended on the emergence of dose-limiting AEs and review of the safety data. Progression to the next higher dose only occurred if the previous dose level was deemed to be safe and well tolerated by the investigator, safety review team, and sponsor. Of the 8 subjects in each cohort, 2 subjects received placebo and 6 subjects received d-methadone.

Subjects were admitted the day prior to receiving the study drug and remained in the clinical research unit (CRU) under clinical supervision for at least 72 hours post-dose. At the discretion of the investigator or designee, the confinement time could have been extended to ensure the safety of each subject. Visits 3 and 4 were follow-up visits approximately 6±2 days and 10±2 days, respectively, after drug administration.

Based on the blinded safety data from Cohorts 1 to 4, single doses of 5 mg, 20 mg, 60 mg, and 100 mg of d-methadone or placebo were well tolerated and there were no dose-limiting AEs.

During all cohorts, subjects were evaluated for safety (AEs, vital signs, electrocardiograms [ECGs], cardiac telemetry, pulse oximetry, clinical laboratory tests), tolerability, and PK. The following signs of opioid toxicity were deemed to be of special interest:

* sustained respiratory depression that results in oxygen saturation below 92%
* QTc prolongation (>500 ms or >70 ms above the baseline)
* protracted nausea and vomiting
* any AE deemed by the investigator to be dose-limiting Safety Analysis Safety and tolerability parameters were listed by treatment and subject and displayed in summary tables using descriptive statistics.

Original terms used to identify AEs were coded using the Medical Dictionary for Regulatory Activities (MedDRA), version 17.1. The number and percentage of subjects with treatment emergent AEs (TEAEs) were summarized by system organ class, preferred term, and treatment and for each treatment by maximum intensity and maximum relationship to study treatment.

Descriptive statistics for vital signs were calculated and presented for each time point by treatment (absolute values and change from baseline). ECG results (absolute values and change from baseline [average of triplicate assessments, where applicable]) were summarized using descriptive statistics; frequencies (numbers and percentages) were calculated for the overall evaluation by scheduled time and treatment. Laboratory data were summarized by the type of test and scheduled visit. Descriptive statistics and number of subjects with laboratory test results below, within, and above normal ranges were tabulated by scheduled time. Abnormal findings in laboratory data were listed with a flag for clinical significance. Medical history abnormalities were coded to MedDRA terms. Physical examination abnormalities were also listed. The original verbatim terms for concomitant medications were coded into drug class and preferred term. These data were listed.

Pharmacokinetic Analysis The PK parameters for d-methadone determined by non-compartmental analysis were summarized by dose. Graphs of concentration (linear and log-linear) vs time were generated. Descriptive statistics were calculated by dose and time point for all d-methadone concentrations. Concentrations below the limit of quantification (BLQ) were set to zero for the generation of summary statistics and mean concentration-time plots.

For the calculation of the PK parameters, concentration-time data were treated as follows: BLQ concentrations prior to the first quantifiable concentration were set to zero; BLQ concentrations after the first quantifiable concentration were treated as missing; pre-dose sampling times relative to dosing were set to zero. Descriptive statistics were calculated by dose. The dose proportionality of Cmax and AUC was assessed by the Hummel method. Tmax and t½ for different doses were compared using the Kruskall-Wallis test to determine whether there was any difference among the treatment groups, and the Wilcoxon rank-sum test for contrasts.

Pharmacodynamic Analysis The PD data at each time point were summarized by descriptive statistics and presented graphically (as appropriate). Derived endpoints were summarized using descriptive statistics.

Outliers were listed by measure and parameter. Pupillometry constriction was listed and grouped by dose and subject with descriptive statistics for changes from baseline for different time points.

ELIGIBILITY:
Inclusion Criteria:

1. healthy male or female subjects, 18 to 55 years of age, inclusive
2. body mass index (BMI) within the range of 18.0 to 30.0 kg/m2, inclusive, and a minimum weight of 50.0 kg
3. non-smoker for at least 3 months and tested negative on a breath carbon monoxide (CO) test
4. male subjects of reproductive potential must have been using and willing to continue using medically acceptable contraception from screening and for at least 2 months after the last study drug administration
5. female subjects of childbearing potential must have been using and willing to continue using medically acceptable contraception for at least 1 month prior to screening (at least 3 months for oral, transdermal, vaginal ring contraceptives) and for at least 2 months after last study drug administration
6. female subjects of non-childbearing potential must have met the criteria defined in the clinical protocol
7. able to speak, read, and understand English sufficiently to allow completion of all study assessments
8. must have understood and provided written informed consent, prior to the initiation of any protocol-specific procedures

Exclusion Criteria:

1. self-reported substance or alcohol dependence (excluding nicotine and caffeine) within the past 2 years, and/or subjects who had ever been in a substance or alcohol rehabilitation program to treat their substance or alcohol dependence
2. subject-reported family history of substance abuse in an immediate family member (i.e., parent, sibling, or child)
3. history or presence of clinically significant abnormality as assessed by physical examination, medical history, 12-lead ECG, vital signs, or laboratory values, which in the opinion of the investigator would jeopardize the safety of the subject or the validity of the study results
4. chronic use of prescribed opioids (i.e., >120 days in a 6-month period) or any recreational use of opioids
5. evidence of clinically significant hepatic or renal impairment, including alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >1.5× upper limit of normal (ULN) or bilirubin >1× ULN
6. history or family history of sudden unexplained death or long QT syndrome
7. QT interval corrected using Fridericia's formula (QTcF) >450 ms in females or >430 ms in males
8. history of hypotension
9. history or presence of any condition in which an opioid was contraindicated (e.g., significant respiratory depression, acute or severe bronchial asthma or hypercarbia, bronchitis, or had/was suspected of having paralytic ileus)
10. history of status asthmaticus, chronic pulmonary disease, or severe allergic reaction (including anaphylaxis) to any substance
11. use of an opioid within the 6 months prior to screening
12. use of a prohibited medication
13. positive urine drug screen
14. positive breath alcohol test; subjects with a positive result may have been rescheduled at the investigator's discretion
15. female subjects who were currently pregnant (had a positive pregnancy test)
16. history of allergy or hypersensitivity to methadone or related drugs (e.g., opioids)
17. positive for hepatitis B, hepatitis C, or human immunodeficiency virus (HIV)
18. donation or loss of more than 500 mL of whole blood within 30 days prior to first drug administration
19. difficulty with venous access or unsuitable or unwilling to undergo catheter insertion
20. treatment with an investigational drug within 5 times the elimination half-life, if known (e.g., a marketed product) or within 30 days (if the elimination half-life is unknown) prior to first drug administration or was concurrently enrolled in any research judged not to be scientifically or medically compatible with this study
21. an employee of the sponsor or research site personnel directly affiliated with this study or their immediate family member, defined as a spouse, parent, sibling, or child, whether biological or legally adopted
22. a subject who, in the opinion of the investigator or designee, was considered unsuitable or unlikely to comply with the study protocol for any reason

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2014-12-04 (Actual); Primary Completion 2015-06-02 (Actual); Study Completion 2015-06-02 (Actual)

PRIMARY OUTCOMES:
Adverse Events (AEs) | Change from pre-dose, 0.5, 1, 2, 3, 5, 8, 12, 24, 36, 48, 60, and 72 hours post-dose, and 7 and 11 days post-dose follow-up
  Spontaneously reported and observed AEs were recorded throughout the study, and AEs were elicited using a non-leading question at designated time points. Regardless of seriousness, intensity, or presumed relationship to study drug, all AEs were recorded in the source documentation from the time of first contact with the subject (e.g., screening) until the end of the follow-up period of the study. AEs that occurred after medical screening and prior to administration of the first dose of study drug were recorded in the source documentation as baseline signs and symptoms.

SECONDARY OUTCOMES:
Plasma levels | Pre-dose, 0.5, 1, 2, 3, 5, 8, 12, 24, 36, 48, 60, and 72 hours post-dose, and 7 and 11 days post-dose follow-up
  Blood samples were collected to determine the plasma levels of d-methadone and l-methadone. The plasma samples were analyzed by the bioanalytical laboratory using validated methods. Plasma samples were shipped frozen on dry ice from the research site to the bioanalytical laboratory.

OTHER OUTCOMES:
Pupillometry | Pre-dose, 0.5, 1, 2, 3, 5, 8, 12, 24, and 48 hours post-dose
  Pupillometry was used as an objective physiological PD measure as it is a sensitive measure of central opioid action and appears to be resistant to tolerance development with repeated administration. An electronic pupillometer was used to measure pupil diameter. Data from a series of frames were used in the calculation, and the final display showed the weighted average and standard deviation of the pupil size. Measurements were collected under mesopic lighting conditions.
Bond-Lader Visual Analog Scale (VAS) | Pre-dose, 0.5, 1, 2, 3, 5, 8, 12, 24, and 48 hours post-dose
  The Bond-Lader Visual Analog Scale (VAS) consists of 16 bi-polar, self-rated, 101-point (from 0 to 100) scales between opposite adjectives. The subjects indicated how they were feeling at the time of assessment. These scales have been shown useful in detecting sedative effects of drugs in normal subjects.
  The 16 scales can be divided into 4 categories of effects, as follows:
  1. Mental sedation or intellectual impairment: Alert/Drowsy, Muzzy/Clear-Headed, Mentally Slow/Quick-Witted, Attentive/Dreamy
  2. Physical sedation or bodily impairment: Strong/Feeble, Well-Coordinated/Clumsy, Lethargic/Energetic, Incompetent/Proficient
  3. Tranquilization or calming effects: Calm/Excited, Contented/Discontented, Troubled/Tranquil, Tense/Relaxed
  4. Other types of feelings or attitudes: Happy/Sad, Antagonistic/Amicable, Interested/Bored, Withdrawn/Gregarious